CLINICAL TRIAL: NCT06852781
Title: Comparison of Spinoglenoid and Suprascapular Notch Approaches and Neuromodulation of the Suprascapular Nerve Under Ultrasonography Guided in Shoulder Pain
Acronym: pain
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: neuromodulation,shoulder pain
Record Dates: First submitted 2025-02-22; First posted 2025-02-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Pain Chronic; Neuromodulation; Ultrasound Guided

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Comparison of Spinoglenoid and Suprascapular Notch Approaches and Neuromodulation of the Suprascapul: Comparison of Spinoglenoid and Suprascapular Notch Approaches and Neuromodulation of the Suprascapular Nerve under Ultrasonography Guided in Shoulder Pain

SUMMARY:
Shoulder pain is a musculoskeletal system (MSS) disease that is frequently seen in adults and tends to become chronic. It ranks 3rd among MSS diseases after low back and knee pain. The main causes of shoulder pain are compression syndromes, acromioclavicular (AC) and glenohumeral joint degeneration, adhesive capsulitis, and biceps tendinopathy. Pathology may be in the joint, bone, muscle, tendon ligament, or bursa. Pain restricts the passive and active range of motion of the shoulder joint, impairing the quality of daily life and activity. It is thought to be between 20% and 50% in the adult population in a 1-year period, and its lifetime prevalence is approximately 10%. Central sensitization develops in cases where the pain is progressive and becomes chronic over time. It has been observed that it becomes chronic in more than 40% of patients in a 1-year period. Thus, shoulder pain becomes a biopsychosocial disease over time.

Physical therapy, medical, interventional methods, and surgery are applied in the treatment of shoulder pain. In physical therapy, exercises and some physical medicine modalities are applied to increase joint range of motion and reduce pain, while in medical treatment, oral analgesics, myorelaxants, and topical analgesics are used. Interventional intra-articular steroid injections and distal suprascapular nerve (SS) blockade radiofrequency applications are among the effective treatment options.

DETAILED DESCRIPTION:
Patients over the age of 18 who have had chronic shoulder pain for more than 3 months, who could not achieve adequate pain palliation despite appropriate medical and physical therapy modalities, and who were treated with SS-PRF between June 2023 and June 2024 with clinical, radiological (MR) and physical examination will be retrospectively screened. The patients whose data can be accessed from the patient file will be recorded for age, gender, body mass index (BMI), duration of symptoms, painful side, pain etiology (subacromial bursitis, impingement syndrome, acromioclavicular degeneration, biceps tendonitis, labral pathologies, shoulder osteoarthritis, etc.), paracetamol dose, and procedure time. Procedure; The patient was taken to the procedure room, monitored [5-lead electrocardiogram (ECG), pulse oximetry, and noninvasive blood pressure], and a vascular access was established in the forearm. After obtaining appropriate sensory and motor responses with a 22 G 100 mm needle and nerve stimulator under ultrasonography guidance, a negative aspiration 5 ml 0.25% bupivacaine diagnostic block was performed with the patient in a semi-sitting position under sterile conditions. In patients who benefited 50% or more from the diagnostic block, a single session of 180 sec, 420 (2 Hz frequency, 45 V, 20 ms) SS-PRF was applied to patients who benefited 50% or more from the diagnostic block with a 100 mm long, 5 mm active tip radiofrequency needle under ultrasonography guidance in a semi-sitting position after obtaining appropriate responses from the suprascapular or spinoglenoid notch (shoulder external rotation and/or abduction).

Geri bildirim gönder Yan paneller Geçmiş Kaydedilenler

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who have pain at or above visual analog scale (VAS) 4 despite pharmacological agents and physical therapy (passive range of motion, strengthening exercises) for more than 3 months and who meet the inclusion criteria will be included in the study.
* Patients with complete data to be scanned in their files

Exclusion Criteria:

* Patients with known malignancy,
* patients who had shoulder injections within the last 3 months,
* patients who changed their medical analgesic treatment or underwent surgery during follow-up,
* patients with previous shoulder surgery or deformity,
* patients with inflammatory arthritis and fibromyalgia,
* patients with known cervical disc herniation,
* patients with pacemakers, pregnant women,
* patients with chronic decompensated disease,
* hemiplegic patients,
* patients with major psychopathology,
* patients allergic to medications used during the procedure,
* patients with infection in the procedure area,
* patients with bleeding disorders, and patients who did not agree to participate in the study were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients over the age of 18 who have pain at or above visual analog scale (VAS) 4 despite pharmacological agents and physical therapy (passive range of motion, strengthening exercises) for more than 3 months and who meet the inclusion criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Activity visual analogue scale (VAS) | one year

CONTACTS AND LOCATIONS:
Overall Officials: altun, Study Director — Kanuni Sultan Süleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided